Calcium Sulfate Spacer in Open Tibia Fractures <a href="NCT03042546">NCT03042546</a> Study name:
ClinicalTrials.gov identifier:
May 1 2016

# Calcium Sulphate Spacer in Open Tibia Fractures with Sub-segmental Bone Loss to Decrease the Need for Secondary Surgery.

HC Sagi, MD

## **Introduction:**

Traumatic tibial shaft fractures can be associated with an increased risk of nonunion and post-traumatic infection/osteomyelitis, particularly when a residual gap exists secondary to bone loss following an open fracture. 1.2 Current recommendations for treatment rely on various strategies involved with aggressive debridement, soft tissue reconstruction, and skeletal stabilization. Initial debridement and early wound management may include the use of antibiotic impregnated poly-methyl-methacrylate (PMMA) beads placed into the bed of the wound to create an antibiotic rich environment in the region of the fracture. 3-5 Subsequent management of the fracture may include sub-acute bone grafting of the bone defect to mitigate the risk of nonunion. Application of Bone Morphogenic Protein-2 (BMP-2) at the time of wound closure and definitive skeletal stabilization has been reported to both decrease the risk of infection and improve union rates. 6 Currently, BMP-2 is approved for use in open tibia factures treated with an intramedullary to decrease both the risk of nonunion and infection – however, BMP-2 can be cost prohibitive and concerns have been raised regarding the potential side effects and complications related to its use. 7

Thus, in order to mitigate the negative financial, medical and social issues associated with infection and nonunion related to open tibia fractures, it is prudent to explore potentially viable alternatives in treating open tibia fractures that may help to decrease the incidence of these sequalae.

One such alternative is the use of Calcium Sulphates (CS) - with or without the addition of antibiotic - in open tibia fractures with boney defects. Calcium Sulphate has been shown to be an effective bone void filler and substitute for autograft in the setting of healing bone defects in a number of animal and human studies.<sup>8-12</sup> Additionally, Calcium sulphate has been shown to be effective both in-vitro and in-vivo as a delivery vehicle for

antibiotics in the setting of treatment for chronic osteomyelitis.<sup>8,13,14</sup> Indeed, in terms of antibiotic elution, it is at least equal to antibiotic laden polymethylmethacrylate (PMMA) in in-vitro studies.<sup>15</sup>

Previously, two retrospective studies on patients with open fractures treated with antibiotic laden Calcium Sulphate have been published on 26 and 15 patients respectively. While the authors were able to demonstrated a union rate of 22/26 and 12/15 respectively, the follow-up was short (10.5 and 8.5 months) and multiple extremity injuries were included in the analysis (such as humerus and metatarsal fractures). The purpose of this study is to prospectively study the effect of antibiotic laden Calcium Sulphate in the acute treatment of open tibia shaft fractures with a boney defect, examining specifically for the need for secondary operation or treatment for infection or nonunion.

### **Methods**:

#### Inclusion Criteria:

- 1. Skeletally Mature
- 2. Open Tibial Shaft Fracture
- **3.** Bone Loss:
  - a. non –segmental bone loss
  - **b.** may require bone grafting
  - c. will not require more than 10cc's of product to fill defect
- 4. Fixation with Intramedullary Rod
- 5. Closeable wound or coverage prior to discharge (2wks max)
- **6.** Radiographic and Clinical Follow-up for one year

#### **Exclusion Criteria:**

- 1. Metabolic Bone Disease
- 2. Immunosuppression
- **3.** Pathological Fracture (Tumor, Pre-existing Infection)
- **4.** Pre-existing Infection
- 5. Soft-tissue coverage not obtained within two weeks from time of injury.
- **6.** Use of Negative Pressure Dressing to definitively manage wound.
- 7. Use of external or implantable bone growth stimulator.
- **8.** Unable to Full Weight Bear immediately post-operative.

#### Data Points:

- 1. Age
- 2. Sex
- 3. Medical Comorbidity
- 4. Smoking Status (Yes or No)
- 5. Wound Size (surface area)
- 6. Wound type (Gustilo Anderson and OTA)
- 7. Number of Surgical Debridements

- 8. Time to definitive closure.
- 9. Soft Tissue Reconstructive Procedure
- 10. Compartment Syndrome (Yes or No)
- 11. Fasciotomy (Yes or No)
- 12. Size of Defect
- 13. Volume of calcium sulphate used
- 14. Treatment of Defect
  - a. Nothing
  - b. PMMA with antibiotic (Vancomycin 1gram + Tobramycin 1gram)
  - c. CS with antibiotic (Vancomycin 1gram + Tobramycin 1gram)
- 15. Need for subsequent secondary treatment:
  - a. Superficial Infection (Antibiotic Treatment)
  - b. Deep Infection (Surgical Treatment)
  - c. Delayed Union (Dynamization, Exchange rodding, Bone grafting)
  - d. Nonunion (Dynamization, Exchange rodding, Bone grafting)

# Methodology:

Patients will be enrolled at a single facility (Harborview Medical Center-HMC). Patients who meet inclusion criteria will be assigned to one of the three treatment groups based on the night of presentation. Currently there are three teams that manage the trauma call at HMC (Red, Green, Blue) and alternate on a strict 1 in 3 rotation schedule. Patients that present on a night when the Red Team is on call will be treated as Group A (Nothing in bone defect at time of closure). Patients that present on a night when the Green Team is on call will be treated as Group B (antibiotic laden PMMA in bone defect at time of closure). Patients that present on a night when the Blue Team is on call will be treated as Group C (antibiotic laden CS in bone defect). All three methods of treatment are considered acceptable current standards of practice in the orthopedic trauma community on a local and national level. All patients will be treated similarly until the time of closure with respect to:

1. Prophylactic Antibiotics administered:

- a. Ancef 1 gram IV q12h until 48 hours following definitive wound closure and final debridement.
- b. Tobramycin 1-2 mg/kg IV q12h until 48 hours following definitive wound closure and final debridement.
- 2. Irrigation and Debridement
- 3. Wound Management
  - a. Clean Type I, II and IIIa wounds will be closed primarily.
  - b. Contaminated Type I, II, and IIIa wounds will be treated with antibiotic bead pouches until closure.
  - c. Type IIIb wounds will be managed with antibiotic bead pouches until flap coverage that will occur no later than one week.

#### 4. Mobilization

a. All patients will be permitted Full Weight Bearing immediately post-operative.

## Risks

There is no risk to the patient as all three treatment methods are current standard of practice both nationally and locally. All patient identifiers will be kept private. All data will be stored on a password protected database available only to the study team.

# **Benefits**

The study performed will provide information regarding the optimal treatment strategy for transverse tibia fractures, and what the expected time to union is when using internal compression. This information is of benefit to patients, particularly when being counseled by surgeons regarding how long they can expect before obtaining radiographic union, and what the potential reoperation rate would be.

# **Procedures to Ensure Confidentiality**

No patient identifiers will be used during the formal study. Identifiers such as name and medical record numbers will be used to identify patients with a transverse tibia fracture, and will be stored on a password protected departmental network in a master file. Data

files will be listed with subject number.

#### **Bibliography:**

- 1) Fong K1, Truong V, Foote CJ, Petrisor B, Williams D, Ristevski B, Sprague S, Bhandari M. Predictors of nonunion and reoperation in patients with fractures of the tibia: an observational study. BMC Musculoskelet Disord. 2013 Mar 22:14:103.
- 2) Schemitsch EH, Bhandari M, Guyatt G, Sanders DW, Swiontkowski M, Tornetta P, Walter SD, Zdero R, Goslings JC, Teague D, Jeray K, McKee MD; Study to Prospectively Evaluate Reamed Intramedullary Nails in Patients with Tibial Fractures (SPRINT) Investigators. Prognostic factors for predicting outcomes after intramedullary nailing of the tibia. J Bone Joint Surg Am. 2012 Oct 3;94(19):1786-93.
- 3) Henry SL1, Ostermann PA, Seligson D. The prophylactic use of antibiotic impregnated beads in open fractures. J Trauma. 1990 Oct;30(10):1231-8.
- 4) Keating JF1, Blachut PA, O'Brien PJ, Meek RN, Broekhuyse H. Reamed nailing of open tibial fractures: does the antibiotic bead pouch reduce the deep infection rate? J Orthop Trauma. 1996;10(5):298-303.
- 5) Moehring HD1, Gravel C, Chapman MW, Olson SA.Comparison of antibiotic beads and intravenous antibiotics in open fractures. Clin Orthop Relat Res. 2000 Mar;(372):254-61.
- 6) Govender S, Csimma C, et al. BMP-2 Evaluation in Surgery for Tibial Trauma (BESTT) Study Group. Recombinant human bone morphogenetic protein-2 for treatment of open tibial fractures: a prospective, controlled, randomized study of four hundred and fifty patients. J Bone Joint Surg Am. 2002 Dec;84-A(12):2123-34.
- 7) Woo EJ1. Adverse events after recombinant human BMP2 in non-spinal orthopaedic procedures. Clin Orthop Relat Res. 2013 May;471(5):1707-11.
- 8) Beuerlein MJ1, McKee MD. Calcium sulfates: what is the evidence? J Orthop Trauma. 2010 Mar;24 Suppl 1:S46-51.
- 9) Elkins AD1, Jones LP. The effects of plaster of Paris and autogenous cancellous bone on the healing of cortical defects in the femurs of dogs. Vet Surg. 1988 MarApr;17(2):71-6.
- 10) Orsini G1, Ricci J, Scarano A, Pecora G, Petrone G, Iezzi G, Piattelli A. Bone-defect healing with calcium-sulfate particles and cement: an experimental study in rabbit. J Biomed Mater Res B Appl Biomater. 2004 Feb 15;68(2):199-208.
- 11) Yang HL1, Zhu XS, Chen L, Chen CM, Mangham DC, Coulton LA, Aiken SS.

- Bone healing response to a synthetic calcium sulfate/ $\beta$ -tricalcium phosphate graft material in a sheep vertebral body defect model. J Biomed Mater Res B Appl Biomater. 2012 Oct;100(7):1911-21.
- 12) Drosos GI1, Ververidis A, Babourda EC, Kakagia D, Verettas DA. Calcium sulfate cement in contained traumatic metaphyseal bone defects. Surg Technol Int. 2012 Dec;22:313-9.
- 13) Fleiter N1, Walter G1, Bösebeck H2, Vogt S2, Büchner H2, Hirschberger W3, Hoffmann R1. Clinical use and safety of a novel gentamicin-releasing resorbable bone graft substitute in the treatment of osteomyelitis/osteitis. Bone Joint Res. 2014 Jul;3(7):223-9.
- 14) Ferguson JY1, Dudareva M, Riley ND, Stubbs D1, Atkins BL2, McNally MA1. The use of a biodegradable antibiotic-loaded calcium sulphate carrier containing tobramycin for the treatment of chronic osteomyelitis: a series of 195 cases. Bone Joint J. 2014 Jun;96-B(6):829-36.
- 15) McConoughey SJ1, Howlin RP, Wiseman J, Stoodley P, Calhoun JH. Comparing PMMA and calcium sulfate as carriers for the local delivery of antibiotics to infected surgical sites. J Biomed Mater Res B Appl Biomater. 2014 Aug 20.
- 16) Cai X1, Han K, Cong X, Cai J, Tong D, Han D, Wang Y, Yu B. The use of calcium sulfate impregnated with vancomycin in the treatment of open fractures of long bones: a preliminary study. Orthopedics. 2010 Mar;33(3).
- 17) Helgeson MD1, Potter BK, Tucker CJ, Frisch HM, Shawen SB. Antibiotic-impregnated calcium sulfate use in combat-related open fractures. Orthopedics. 2009 May;32(5):323.
- 18) Borrelli J Jr1, Prickett WD, Ricci WM. Treatment of nonunions and osseous defects with bone graft and calcium sulfate. Clin Orthop Relat Res. 2003 Jun;(411):245-54.